CLINICAL TRIAL: NCT04703777
Title: Retrospective Study on the Relationship Between Social Status and Use of Healthcare Services During the Confinement Period Linked to the COVID-19 Epidemic in Bas-Rhin, France
Brief Title: Relationship Between Social Status and Use of Healthcare Services During the Confinement Period Linked to the COVID-19 Epidemic
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7814
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-01

CONDITIONS: Covid-19
Keywords: COVID-19; Coronavirus; Sars-cov-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemics have always affected the most disadvantaged social categories more intensely. This social inequality is expressed in the use of care and emergencies: greater frequency but also greater seriousness. Our hypothesis is that, during a period of confinement, the most disadvantaged populations are more affected by the COVID-19 infection than the rest of the population. The number of remedies is greater, as is the severity of the forms of infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or over
* Calling center 15 from March 17 at noon and until the end of the confinement period (May 31, 2020) for one of the following reasons that may be related to COVID-19: cough, fever, rhinitis, diarrhea, pain thoracic, odynophagia, diarrhea, anosmia, ageusia, whose calling address belongs to Bas-Rhin Or
* Supported (consultation or hospitalization) at the HUS for a COVID-19 infection and included in the COVID-HUS base and residing in the Bas-Rhin.

Exclusion Criteria:

* Patient under the protection of justice
* Patient under guardianship, curatorship
* Patient taken care of at the screening center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient suspected of covid-19
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-04-04 (Actual)

PRIMARY OUTCOMES:
Retrospective study on the relationship between social status and use of healthcare services during the confinement period linked to the COVID-19 epidemic in Bas-Rhin, France | Files analysed retrospectily from March 17, 2020 to May 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu OBERLIN, Study Director — Adult Emergency Department - Strasbourg University Hospitals
Locations (1):
- Adult Emergency Department - Strasbourg University Hospitals, Strasbourg, France